CLINICAL TRIAL: NCT02996604
Title: Acupuncture for Functional Dyspepsia: a Functional Magnetic Resonance Imaging (fMRI) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15QNJJ0008; 81473602 (Other Grant/Funding Number: National Scientific Foundation Committee of China)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Functional Dyspepsia
Keywords: acupuncture; functional dyspepsia; functional magnetic resonance imaging (fMRI)
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Low-He point(ST36) (Experimental): Zusanli (ST36, the Low-He point of stomach) is the most important point for gastrointestinal disorder, including functional dyspepsia. Everyone in the group will be punctured at unilateral Zusanli.
  Interventions: Other: acupuncture
- Mu point(CV12) (Experimental): Zhongwan (CV12, the Mu point of stomach) is also good at regulating gastric function. Everyone in the group will be punctured at Zhongwan.
  Interventions: Other: acupuncture
- He-Mu-point combination(ST36 and CV12) (Active Comparator): In traditional Chinese acupuncture theory，synergistic effect can be produced by acupoints combination and the He-Mu-point combination is a classical acupoints combination formula for gastrointestinal diseases. Everyone in the group will be punctured at unilateral Zusanli and Zhongwan.
  Interventions: Other: acupuncture

INTERVENTIONS:
Other: acupuncture — Manual acupuncture treatment will be conducted. thirty minutes duration every time, five times per week for one course, a total four courses.
  Other Names: Manual acupuncture

SUMMARY:
He-Mu-point combination（ST36 and CV12） is one of the most commonly used acupoints combination with synergistic effect for functional dyspepsia(FD). The investigators design the trial to identify the efficacy and explore the central integrated mechanism of puncturing at He-Mu-point combination on FD with functional magnetic resonance imaging (fMRI).

DETAILED DESCRIPTION:
105 participants with functional dyspepsia will be allocated into three groups: Low-He point group, Mu point group and He-Mu-point combination group.Every participant will receive 20 sessions of manual acupuncture treatment during 4 weeks. Clinical evaluations will be assessed three times, as measured after randomization, 10 and 20 sessions of treatment.The fMRI scans will be conducted twice, after randomization and treatment completion.

ELIGIBILITY:
Inclusion Criteria:

1. right handed，age between 18 and 45 years old, college degree or above;
2. match the Rome III criteria on FD;
3. no local organic disease by gastroscope examination;
4. before entering the study, without taking any prokinetic agents at least 15days and participating in other clinical study;
5. signing an informed consent in writing by the participant or the immediate family member.

Exclusion Criteria:

1. consciousness, cannot express subjective symptoms and psychiatric participants;
2. participants with advanced cancer or other serious wasting diseases, easy to be infected and bleeding;
3. complicating with severe cardiovascular, hepatic,nephritic,digestive, hematopoietic system diseases;
4. impregnate or lactation female;
5. severe depression and anxiety symptoms;
6. female with serious dysmenorrhea;
7. obvious headache, migraine, history of head injury.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Nepean Dyspepsia Index (NDI) | 4 weeks after allocation

SECONDARY OUTCOMES:
Self-Rating Anxiety Scale | 0 day,2, 4weeks after allocation
Self-Rating Depression Scale | 0 day,2, 4weeks after allocation
Leeds dyspepsia questionnaire | 0 day,4 weeks after allocation
brain MRI data | 0 day,4weeks after allocation
The incidence of adverse events during the 4 weeks | 4weeks after allocation

CONTACTS AND LOCATIONS:
Overall Officials: Fang Zeng, professor, Study Chair — Chengdu University of Traditional Chinese Medicine
Locations (1):
- Chengdu University of Traditional Chinese Medicine, Chengdu, Sichuan, China